CLINICAL TRIAL: NCT02781753
Title: A Phase 1 Study to Evaluate the Pharmacokinetic and Pharmacodynamic Profile, Safety, and Tolerability of Escalating Single Dose Recombinant Human Serum Albumin/Interferon alpha2b Fusion Protein in Healthy Chinese Volunteers
Brief Title: Study of Recombinant Human Serum Albumin/Interferon alpha2b Fusion Protein in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 921601
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — Serum Albumin, Human; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Serum Albumin/interferon alpha2b (Experimental): Human Serum Albumin/interferon alpha2b fusion protein 300-1200 μg single dose S.C.
  Interventions: Biological: Human Serum Albumin/interferon alpha2b
- Pegasys (Active Comparator): Peginterferon 180 μg single dose S.C.
  Interventions: Biological: Peginterferon 180 μg single dose S.C.

INTERVENTIONS:
Biological: Human Serum Albumin/interferon alpha2b — Human Serum Albumin/interferon alpha2b fusion protein 300-1200 μg single dose S.C. at Day0
  Arms: Human Serum Albumin/interferon alpha2b
Biological: Peginterferon 180 μg single dose S.C. — Pegasys 180 mcg S.C. single dose on Day 0
  Arms: Pegasys

SUMMARY:
The purpose of this study is to evaluate the dosages of recombinant human serum albumin/interferon alpha2b fusion protein injection in healthy subjects.

DETAILED DESCRIPTION:
This is an open-label study that will be conducted at a single site in China to characterize the PK/PD profile, safety and tolerability of Recombinant Human Serum Albumin/interferon alpha2b Fusion Protein in healthy subjects. Subjects will receive a single dose of Recombinant Human Serum Albumin/interferon alpha2b Fusion Protein or active comparator Pegasys at Day 0. The total duration of study participation is up to 6 weeks for each subject. Subjects will complete a follow-up visit at Day 28 after the dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy males or females between 18 to 45 years old, inclusive
* Must have a body mass index (BMI) of 19 to 25 kg/m2, inclusive, and a minimum body weight of 50.0 kg

Exclusion Criteria:

* History of any clinically significant laboratory abnormalities, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major diseases
* Female subjects who are pregnant or breastfeeding
* Any previous treatment with Human Albumin Interferon fusion protein

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events after single dose | 4 weeks
  Frequency and severity of all adverse events on the part of the participants, including frequency and severity of drug-related adverse events.

SECONDARY OUTCOMES:
Pharmacokinetics of interferon after single dose | 4 weeks
  Peak plasma concentration(Cmax)
Pharmacokinetics of interferon after single dose | 4 weeks
  Area under the plasma concentration versus time curve (AUC)
Plasma concentration of Neopterin after single dose | 4 weeks
  Plasma concentration of Neopterin after single dose
Pharmacokinetics of interferon after single dose | 4 weeks
  Peak time(Tmax)
Pharmacokinetics of interferon after single dose | 4 weeks
  Half-life period(T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Meixia Wang, Professor, Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No